CLINICAL TRIAL: NCT01846221
Title: Comparison of Fentanyl-bupivacaine and Clonidine-bupivacaine for Breakthrough Pain in Advanced Labor in Patients With Continuous Epidural Analgesia
Brief Title: Comparison of Epidural Fentanyl and Clonidine for Breakthrough Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Allison Lee, Assistant Professor of Clinical Anesthesiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAL4101
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Results first posted 2018-05-03 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Labor Pain
Keywords: Analgesia; Epidural; Pregnancy; Labor; Clonidine; Fentanyl; Bupivacaine; Childbirth
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Clonidine; Fentanyl

STUDY DESIGN:
Intervention Model Description: Subjects will randomly receive either a mixture of 100 mcg of clonidine and 12.5 mg of bupivacaine for a total volume of 10 ml ("CLON" group) and the other group will receive 100 mcg of fentanyl and 12.5 mg of bupivacaine for a total volume of 10 ml ("FENT" group). If the treatment is declared a failure, the patient will receive the alternative of the initial treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Group assignment will be performed by opening a previously prepared numbered opaque envelope containing the assignment "CLO" or "FENT". The investigator preparing the study drug will not reveal the group assignment. The investigator administering the drug (different from the investigator preparing the drug) and assessing the outcomes will be blinded to the group assignment. The participant will also be blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clonidine (Experimental): Participants randomized to this arm of the study receive 100 micrograms clonidine with the bupivacaine in their epidural when requesting pain relief in advanced labor
  Interventions: Drug: Clonidine
- Fentanyl (Experimental): Participants randomized to this arm of study will receive 100 mcg fentanyl with the bupivacaine in their epidural when requesting pain relief in advanced labor
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Clonidine — Subjects randomized to clonidine will receive a mixture of 100 micrograms clonidine and 12.5 mg bupivacaine 10 ml of volume.
  Other Names: DuraClon
  Arms: Clonidine
Drug: Fentanyl — Subjects randomized to fentanyl will receive 100 mcg fentanyl and 12.5 mg bupivacaine in 10 ml of volume.
  Other Names: Sublimaze
  Arms: Fentanyl

SUMMARY:
Epidural analgesia has proven to be an effective method for severe pain relief associated with labor and delivery. During labor, a low dose continuous infusion of local anesthetic and narcotic will be administered through an epidural catheter. As labor progresses and the baby's head makes it way through the pelvis, breakthrough pain may emerge and often needs further treatment. The investigators provide pain relief by administering analgesics through the epidural catheter. The patients will be randomly assigned to receive one of two medication mixtures believed to be successful in treating this type of pain associated with advanced labor. After this initial treatment, if pain relief is not attained, the patient may receive the other medication as well. The medications used in this study have been used at this institution for some time and have been found to be safe for mother and baby. The opioid (fentanyl) dose is small and only a small fraction will be transmitted to the baby. The other medication (clonidine) better known as a blood pressure medication has also been used for pain relief. Studies and clinical experience have shown that clonidine when given epidurally in the doses used in this study has minimal, if any effect, on the blood pressure of the mother or of the baby. The investigators will record medical and obstetric history and labor progress relevant to the patient. The patient will be asked questions regarding labor pain and side effects before and after the analgesic is administered. The primary objective is to determine which treatment regimen is more successful in abolishing breakthrough pain in advanced labor.

DETAILED DESCRIPTION:
Epidural analgesia is a popular choice among patients for relief of severe pain associated with labor and delivery. Currently, at the investigators' institution the investigators use a continuous infusion of low dose local anesthetic and narcotic (12 ml/hr of 0.0625% bupivacaine with 2 micrograms/ml fentanyl) after the initial spinal or epidural dose to maintain patient comfort until delivery. This dose of the infusion is chosen because it often provides adequate comfort without interfering with the mobility of the patient and her ability to effectively push during delivery. However, this low-dose epidural infusion strategy often results in recurrence of pain after an initial pain-free period. This recurring pain is known as breakthrough pain and is alleviated by administering small boluses of analgesics via the epidural catheter.

The pain occurring in labor is initially of visceral origin and is mediated by pain fibers originating from the low thoracic and upper lumbar segments of the spinal cord. As labor progresses to the late first phase (also known as transitional stage), pain sensations originating from the distension of the pelvic floor, vagina and perineum adds a somatic component to labor pain. This type of breakthrough pain, mediated by nerve fibers originating from the sacral nerves at dermatomes S2-S4, is often difficult to treat. Patients may experience inadequate analgesia even after boluses of analgesics are administered. Inadequate analgesia is deleterious due to subjective discomfort with its associated neurohumoral and physiological changes, and can be an initiator of the urge to bear down (push). Pushing before complete dilation of the cervix may lead to swelling, cervical injury and premature exhaustion of the mother. Adequate pain control will allow the cervix to fully dilate and motivate the mother to push effectively at the appropriate time. Although requests from patients to alleviate late stage breakthrough pain are common, there are no established data in the literature regarding the most effective strategy for pain management in this stage of labor.

This study is designed to compare the efficacy of two treatments for controlling late first stage breakthrough pain during labor: clonidine-bupivacaine versus fentanyl-bupivacaine. Both strategies are used at Columbia University Medical Center (CUMC) in this clinical situation, and there is no clear evidence whether one is superior.

ELIGIBILITY:
Inclusion Criteria:

* women in labor at term pregnancy
* healthy
* epidural analgesia in place
* breakthrough pain in advanced labor

Exclusion Criteria:

* chronic pain syndrome
* receiving systemic opioids within 4 hours
* receiving chronic antidepressants, clonidine, opioids

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-07-15 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Lee, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The Journal of the American Society of Anesthesiologists Abstract — http://www.asaabstracts.com/strands/asaabstracts/abstract.htm?year=2017&index=14&absnum=4456

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clonidine | Fentanyl
Started | 50 | 51
Completed | 47 | 51
Not Completed | 3 | 0
Not completed — Catheter Failure | 2 | 0
Not completed — Age Exclusion | 1 | 0

BASELINE CHARACTERISTICS:
Population: 3 subjects in the Clonidine group were not included in the analysis due to the following reasons: 2 catheter failures, 1 age limit exclusion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clonidine | Fentanyl | Total
Number analyzed (Participants) | 47 | 51 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 51 | 98
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 51 | 98
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 10 | 26
  White | 27 | 31 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 7 | 8
Region of Enrollment [Number; unit: participants]
  United States | 47 | 51 | 98

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Success Rate at 15 Minutes Post-epidural Bolus Injection
Description: Pain Visual Analogue Scale (VAS) was evaluated every 5 min for 15 min. 'Success' is defined as at least a 4-point reduction in VAS at 15 min. (0=no pain, 10= worst pain)
Time Frame: Baseline, 15 Minutes post epidural administration
Population: 3 subjects in the Clonidine group were not included in the analysis due to the following reasons: 2 catheter failures, 1 age exclusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Clonidine | Fentanyl
Number analyzed (Participants) | 47 | 51
Participants | 31 | 38
Statistical Analysis 1: Comparison: Clonidine vs Fentanyl; Test type: Other; p = 0.38, ANOVA

2. Secondary Outcome: Maternal Systolic Blood Pressure
Description: Blood pressure will be measured at different timepoints.
Time Frame: Baseline, 30 Minutes post epidural administration
Population: 46 out of 47 participants were included from the Clonidine group due to 1 participant did not have blood pressure taken at 30 minutes. 48 out of 51 participants were included from the Fentanyl group due to 3 participants did not have blood pressure taken at 30 minutes.
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | Clonidine | Fentanyl
Number analyzed (Participants) | 46 | 48
mm Hg
  Baseline | 123 [91 to 172] | 121 [83 to 146]
  30 Minutes | 116 [87 to 150] | 118 [87 to 141]

3. Secondary Outcome: Maternal Heart Rate
Description: Heart rate will be measured at different timepoints.
Time Frame: Baseline, 30 Minutes post epidural administration
Population: 48 out of 51 participants were included from the Fentanyl group due to 4 participants did not have heart rate taken at 30 minutes.
Measure: Mean (Full Range); unit: beats per minute (BPM)
Arm/Group | Clonidine | Fentanyl
Number analyzed (Participants) | 47 | 48
beats per minute (BPM)
  Baseline | 87 [57 to 155] | 84 [65 to 113]
  30 Minutes | 84 [54 to 131] | 85 [62 to 112]

4. Secondary Outcome: Neonatal Apgar Score
Description: The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health.
Time Frame: 1 minute and 5 minutes post delivery
Measure: Mean (Full Range); unit: Apgar score
Arm/Group | Clonidine | Fentanyl
Number analyzed (Participants) | 47 | 51
Apgar score
  1 Minute | 8.53 [6 to 9] | 8.24 [1 to 9]
  5 Minutes | 8.94 [8 to 9] | 8.88 [6 to 9]

5. Secondary Outcome: Number of Spontaneous Vaginal Deliveries
Description: Mode of delivery: spontaneous vaginal or instrumental vaginal versus cesarean.
Time Frame: Upon delivery (approximately up to 8 hours from baseline)
Measure: Number; unit: spontaneous vaginal deliveries
Arm/Group | Clonidine | Fentanyl
Number analyzed (Participants) | 47 | 51
spontaneous vaginal deliveries | 38 | 40

ADVERSE EVENTS:
Time Frame: Up to 2 hours after initial epidural bolus (study drug) injection
Arm/Group | Clonidine | Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/51
Other Adverse Events (participants affected / at risk) | 0/47 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT01846221/Prot_SAP_000.pdf